CLINICAL TRIAL: NCT03689842
Title: Feasibility Study of Uterine Transplantation From Living Donors in Terms of Efficacy and Safety in Patients With Mayer-Rokitansky-Küster-Hauser Syndrome (MRKH)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/26
Record Dates: First submitted 2018-07-13; First posted 2018-09-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Mayer Rokitansky Kuster Hauser Syndrome
MeSH Terms: conditions — Mullerian aplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Couple donor - recipient (Experimental)
  Interventions: Procedure: Uterine transplantation

INTERVENTIONS:
Procedure: Uterine transplantation — Uterine transplantation from living donor

SUMMARY:
In France, one in 4500 women is affected by the MayerRokitantskyKüsterHauser (MRKH) syndrome which is characterized by the absence of uterus at birth. Currently, the only solutions for these patients are:

* Gestational surrogacy, prohibited in France
* Adoption
* Resignation

Uterine transplantation could become a good alternative.

This study is conducted in 10 patients with MRKH type I syndrome, who will be transplanted from a living donor uterus

DETAILED DESCRIPTION:
The aim of the study is to obtain a pregnancy after uterine transplantation from a living donor. Also, this study will assess (anatomically and functionally) the issue of the transplants of a uterus taken from a living donor and the safety of the living donor (functionally and psychologically)

ELIGIBILITY:
Inclusion Criteria:

Graft recipient is a patient with Mayer-Rokitansky-Küster-Hauser Type I Uterine Vaginal Agenesis (without renal, cardiac and bone malformations):

* Being aged between 18 and 38 years old
* In stable couple, with a pregnancy project, favorable psychological evaluation
* No history of cancer and transfusion

The living donor is a woman related to the Graft recipient with

* Absence of comorbidity (neurological, nephro-urological pathology, infectious, psychiatric or psychological pathology)
* Absence of uterine surgery, abdomino-pelvic major pathology history

Exclusion Criteria:

Graft recipient:

* Extreme oligo-astheno-spermia and azoospermia in the husband
* History of abdominopelvic surgery excluding uncomplicated appendectomy; vaginal residue not allowing anastomosis

Living donor :

* Known thromboembolic risk factor
* No Compatibility with the recipient (group, rhesus, HLA)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2027-12-14 (Estimated); Study Completion 2034-12-14 (Estimated)

PRIMARY OUTCOMES:
Pregnancy | 3 years
  Obtaining of a pregnancy after uterine transplantation from a living donor

SECONDARY OUTCOMES:
Safety assessment of the donor, the recipient and the fœtus | 7 years
  Monitoring of all the Adverse events
Psychological assessment of the donor and the recipient | 7 years
  Psychological consequences linked to the procedure determined by repeated interviews with psychologists
Graft Rejection assessment | 5 years
  Donor-specific antobodies monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goetgheluck J, Carbonnel M, Ayoubi JM. Robotically assisted gynecologic surgery: 2-year experience in the French foch hospital. Front Surg. 2014 May 5;1:8. doi: 10.3389/fsurg.2014.00008. eCollection 2014. PMID 25593933
- [Background] Brannstrom M, Johannesson L, Bokstrom H, Kvarnstrom N, Molne J, Dahm-Kahler P, Enskog A, Milenkovic M, Ekberg J, Diaz-Garcia C, Gabel M, Hanafy A, Hagberg H, Olausson M, Nilsson L. Livebirth after uterus transplantation. Lancet. 2015 Feb 14;385(9968):607-616. doi: 10.1016/S0140-6736(14)61728-1. Epub 2014 Oct 6. PMID 25301505
- [Background] Carbonnel M, Abbou H, N'guyen HT, Roy S, Hamdi G, Jnifen A, Ayoubi JM. Robotically Assisted Hysterectomy versus Vaginal Hysterectomy for Benign Disease: A Prospective Study. Minim Invasive Surg. 2013;2013:429105. doi: 10.1155/2013/429105. Epub 2013 Jul 7. PMID 23936645
- [Background] Gauthier T, Lavoue V, Piver P, Aubard Y, Ayoubi JM, Garbin O, Agostini A, Collinet P, Morcel K; Comite d'etude de la Transplantation Uterine en France (CETUF) du CNGOF. Which neovagina reconstruction procedure for women with Mayer-Rokitansky-Kuster-Hauser syndrome in the uterus transplantation era? Editorial from the French Uterus Transplantation Committee (CETUF) of CNGOF. J Gynecol Obstet Hum Reprod. 2018 Apr;47(4):175-176. doi: 10.1016/j.jogoh.2018.01.003. Epub 2018 Jan 31. No abstract available. PMID 29391294
- [Background] Grynberg M, Ayoubi JM, Bulletti C, Frydman R, Fanchin R. Uterine transplantation: a promising surrogate to surrogacy? Ann N Y Acad Sci. 2011 Mar;1221:47-53. doi: 10.1111/j.1749-6632.2011.05952.x. PMID 21401629